CLINICAL TRIAL: NCT06065488
Title: Functional Ankle Taping Correction on Plantar Foot Ulcer Healing in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, lectrurer of physical therapy for general surgery and dermatology,MTI University, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004688
Record Dates: First submitted 2023-09-20; First posted 2023-10-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Foot Ulcer
Keywords: plantar foot ulcers; ankle kinesiotap; wound healing; chronic wounds; diabetic patients
MeSH Terms: conditions — Foot Ulcer

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1.Group A (Ankle KT group): (Experimental): This group includes 35 patients with chronic unhealed plantar foot ulcers for longer than three months; they will receive functional ankle taping, medical treatment, and dressing according their cases. The tape was applied for 5 days and then removed for 1 day to allow skin perspiration. This process was repeated for successive 8 weeks. The patient was instructed to avoid vigorous activities for 30 min, which is required for the glue to become fully activated (Andrýsková et al., 2020)
  Interventions: Device: ankle kinesio tap
- 2.Group B (Control group Ankle shame KT ): (Sham Comparator): This group includes 35 patients with chronic unhealed plantar foot ulcers for longer than three months. Shame taping group, a placebo taping method considered to be ineffective ( not from insertion to origin of muscles) with the same material without tension , they will receive medical treatment, and dressing according their cases The shame tape was applied for 5 days and then removed for 1 day to allow skin perspiration. This process was repeated for successive 8 weeks. The patient was instructed to avoid vigorous activities for 30 min, which is required for the glue to become fully activated. (Andrýsková et al., 2020)
  Interventions: Device: ankle kinesio tap

INTERVENTIONS:
Device: ankle kinesio tap — Kinesio Tape is popular among athletes and non-athletes for its ability to protect, support, and promote activity in overworked muscles. Few people are aware, however, that its healing benefits don't end there. Research studies show that taping ankle with Kinesio Tape actually improves ankle range of motion.

SUMMARY:
This study will investigate the effects of Functional ankle taping correction on plantar foot ulcer healing in diabetic patients. This study will be carried out at the outpatient clinic of the faculty of physical therapy, modern university for technology and information, Om El masryeen general Hospital and El Rahma - private clinic.

All participants will sign a written consent form after receiving full information about the purpose of the study, procedure, possible benefits, privacy, and use of data.

DETAILED DESCRIPTION:
Design of the study: Randomized controlled trial.

Subject's selection:

Estimated sample size is 70 subjects the actual sample size will be calculated after pilot study. They will be assigned into two equal groups:

1. Group A (Ankle KT group):

   This group includes 35 patients with chronic unhealed plantar foot ulcers for longer than three months; they will receive functional ankle taping, medical treatment, and dressing according their cases. The tape was applied for 5 days and then removed for 1 day to allow skin perspiration. This process was repeated for successive 8 weeks. The patient was instructed to avoid vigorous activities for 30 min, which is required for the glue to become fully activated (Andrýsková et al., 2020)
2. Group B (Control group Ankle shame KT ):

This group includes 35 patients with chronic unhealed plantar foot ulcers for longer than three months. Shame taping group, a placebo taping method considered to be ineffective ( not from insertion to origin of muscles) with the same material without tension , they will receive medical treatment, and dressing according their cases The shame tape was applied for 5 days and then removed for 1 day to allow skin perspiration. This process was repeated for successive 8 weeks. The patient was instructed to avoid vigorous activities for 30 min, which is required for the glue to become fully activated. (Andrýsková et al., 2020) Patients were followed for 8 weeks or until ulcer healing, whichever came first. The protocol was designed according to the fundamental treatment principal of the expert panel to the 2022 American Diabetic Association consensus development conference on diabetic foot wound care.

ELIGIBILITY:
1. Inclusion Criteria:

   The subject selection will be according to the following criteria:
   * Undergoing treatment for a Wagner grade II or III diabetic foot ulcer
   * Age between 42 and 60 years.
   * No systemic diseases such as musculoskeletal disorders, heart diseases, or neurological diseases that can hinder ability to participate in the study
   * Not receiving other treatments that could affect wound healing (negative-pressure wound treatment, hyperbaric oxygen treatment, a special wound care product, special wound dressing, or growth factor.
   * Not using another complementary treatment method (herbal wound care products and Participating subjects were required to be able to walk 10 m unassisted.
   * Absence of protective sensation on the plantar foot as determined using a 10-gram monofilament following criteria from the International Working Group on the Diabetic Foot 2023
   * All the patients have active unilateral plantar DFU at least 1cm2 (greatest length x greatest width) and not healed > 3months duration.

   Never received the same intervention from other researchers and health Professionals..

   • Ability to walk independently for 30 steps or 10 min.
2. Exclusion Criteria:

The potential participants will be excluded if they meet one of the following criteria:

* Patients with inadequate vascular circulation (ankle-brachial pressure index <0.8 or toe systolic blood pressure <40 mmHg)
* Patient with skin allergy with generalized osteoporosis, or who had fractures of any bones in the lower extremity.
* Previous ankle pathology or surgery to the lower limb within the last 12 months, current illness or infection, neurological deficits affecting the lower limb and skin conditions or edema affecting the lower limb ,Severe uncontrolled hypertension.
* Pregnant women.
* Un controlled diabetes
* Pedal amputations and arthritis.
* Ulcer developed secondary to acute trauma; ulcer developed secondary to burns.
* Foot deformities included hallux valgus, hallux rigidus, pes planus, pes cavus, low forefoot arch, and hammer toes, Skin callosities, heel fissures, a hypotrophic fat pad, and nail deformities

Ages: 42 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Maximum plantar peak pressures of ulcerated foot | Baseline then after 8 weeks
  Maximum plantar peak pressures were measured using Tekscan® pressure mat system (Boston , MA). - Patients were given time to familiarise themselves with the protocol. - Prior to testing he mat was calibrated for each individual's mass using mat-Scan® System Research software (Tekscan, Boston, MA). - Once calibration was completed Patient was asked to walk across the plantar pressure mat which placed in the center of walkway - The method has been previously validated and involves each participant taking two steps before landing on the pressure mat. - Trials were excluded and repeated if a participant appeared to target the platform and alter their gait pattern to ensure full contact with the mat - - Collecting data from mat-based Stride way System, a 150 cm long and 60 cm Wide to generate maximum Peake pressure by quantifying the pressure exerted on the force sensors\ - Direct cont

SECONDARY OUTCOMES:
Ankle dorsiflexion range of motion of ulcerated foot | Baseline then after 8 weeks
  The maximum dorsiflexion angle at the ankle joint was measured with hand - held standard goniometer in a standing position with the knee extended, with the heel in contact with the ground. Participants were asked to lean forward, directing their knees toward the wall. While the participant maintained his or her maximal dorsiflexion position, a standard goniometer was aligned with floor (stable arm) and through the shaft of the fibula (mobile arm) by visually bisecting the lateral malleolus and the fibular head. Participants were allowed three practice trials.
Wound surface area by +Wound Desk mobile application | Baseline then after 8 weeks
  To start working with the application, it is required to sign in into the account. A patient's profile is completed; where it is required to indicate the location and how the trauma happened (one of several options is offered). Based on the completed profile of the dynamic monitoring process, one of standard treatment options is offered. To obtain photos, Take anew photo mode is selected in the application, which turns on the mobile application photo camera. +WD indicator should be placed next to the studied wound. The wound area is photographed, and the program recognizes +WD marker thereafter and requires a manual detection of wound borders using a thumb knob. Next, an automatic calculation of the wound surface area is performed and the result is provided
Wound volume assessment | Baseline then after 8 weeks
  - Using sterilized siring and saline solution. - Filing the sterilized siring of 5 cm3 with saline solution. - Then filing the wound by the kwon volume of the saline solution - It is an easy accurate method for wound volume estimation

CONTACTS AND LOCATIONS:
Overall Officials: El fahl, ph.d, Study Chair — faculty of physical therapy .Modern university for information and technology
Locations (1):
- Ahmed Mohamed Ahmed Abdelhady, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bus SA, van Deursen RW, Armstrong DG, Lewis JE, Caravaggi CF, Cavanagh PR; International Working Group on the Diabetic Foot. Footwear and offloading interventions to prevent and heal foot ulcers and reduce plantar pressure in patients with diabetes: a systematic review. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:99-118. doi: 10.1002/dmrr.2702. PMID 26342178
- [Background] Lazzarini PA, Jarl G, Gooday C, Viswanathan V, Caravaggi CF, Armstrong DG, Bus SA. Effectiveness of offloading interventions to heal foot ulcers in persons with diabetes: a systematic review. Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1(Suppl 1):e3275. doi: 10.1002/dmrr.3275. PMID 32176438
- See also: Effectiveness of offloading interventions to heal foot ulcers in persons with diabetes: a systematic review — https://pubmed.ncbi.nlm.nih.gov/?term=effectiveness+of+offloading+interventions+to+heal+foot+ulcer+in+persons+with+diabetes%3A+a+systematic+review